CLINICAL TRIAL: NCT05820386
Title: Assessment of Skin-to-skin Contact During the Transfer of Very Preterm Infants From the Delivery Room to the Neonatal Intensive Care Unit : a Randomised Controlled, Non-inferiority, Open-label Trial, in Comparison With Transfer in Incubator
Brief Title: Skin-to-skin Contact During the Transfer From the Delivery Room to the Neonatal Intensive Care Unit: Impact on Very Preterm Infants and Their Parents
Acronym: TRANSPAPNEO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DR210297
Record Dates: First submitted 2023-03-23; First posted 2023-04-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Skin to Skin; Premature Newborns
Keywords: Skin to skin; Premature newborns
MeSH Terms: interventions — Incubators

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skin-to-skin contact during the transfer between the delivery room and the neonatal care unit (Experimental): Preterm infants will be transferred using a direct skin-to-skin contact with their father from the delivery room to the intensive neonatal care.
  Interventions: Procedure: Skin-to-skin Contact (SSC)
- Transfer in incubator between the delivery room and the neonatal care unit (Active Comparator): Preterm infants will be transferred in an incubator set to 36°C from the delivery room to the intensive neonatal care.
  Interventions: Procedure: Incubator

INTERVENTIONS:
Procedure: Skin-to-skin Contact (SSC) — For the Skin-to-skin Contact (SSC) transfer, the bare-chested father will seat in a wheelchair. Newborns who will wear only a diaper and a cotton cap or noninvasive ventilation headgear will be placed in the kangaroo position against the father's chest to ensure direct contact with the father's skin. Preterm infants with gestational age less than 33 weeks will be wrapped with their father using plastic bags plus warmed cotton towels. More gestationally mature infants will be wrapped with only warmed cotton wraps. The newborn's heart rate, oxygen saturation and skin temperature will be monitored throughout the procedure.
  Arms: Skin-to-skin contact during the transfer between the delivery room and the neonatal care unit
Procedure: Incubator — In the incubator group, infants will be transferred after resuscitation in an incubator with air temperature set to 36°C. The newborn will be laid on his/her back in a polyethylene bag with a cap. The newborn's heart rate, oxygen saturation and skin temperature will be monitored throughout the procedure.
  Arms: Transfer in incubator between the delivery room and the neonatal care unit

SUMMARY:
Developmental care are recognized as a standard of care for preterm infants in neonatal intensive care units. Regular skin-to skin contacts during the neonatal stay show short and long-term beneficial effects on preterm infants and their parents. Skin-to-skin contact provides hemodynamic and thermal stability in preterm infants. Regarding parents, skin-to-skin contact sustains the parental bonding, and reduces stress and anxiety related to hospitalization. As a result, early skin-to-skin contact has been associated with an improvement of neurological outcome in very preterm infants.

Thermal stability is crucial during the first hour of life in preterm infants. A temperature at admission in the neonatal intensive care unit below 36.5°C or above 37.2°C has been associated with an increase in neonatal morbidity and mortality.

Early skin-to-skin contact between a newborn and his/her mother in the delivery room significantly decreases the occurrence of hypothermia below 35.5°C.

The practice of skin-to-skin transfer from the delivery room is emerging in France. Pilot studies have been carried out by French neonatal teams that showed the feasibility of this practice in late-preterm, near-term and term infants. Although skin-to-skin contact routinely involves very preterm infants in neonatal intensive care units worldwide, the feasibility and safety of skin-to-skin contact during the transfer from delivery room to the neonatal unit is poorly documented in very preterm infants. Previous data of our team showed that transfer of preterm infants with non-invasive ventilation using skin-to-skin contact was feasible and safe but concerns emerged about the thermal conservation during the procedure.

The main hypothesis of this study is that skin-to skin contact during the transfer from the delivery room to the neonatal intensive care unit could prevent heat losses in preterm infants as well as the transfer in incubator. Another hypothesis is that very early skin-to-skin contact could positively influence the neonatal course and the parental experience in the neonatal care unit.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age < 34 weeks
* Singleton pregnancy
* Inborn birth, i.e., in the maternity ward of investigating centres
* Need of hospitalization in the neonatal intensive care unit
* Oral and written information of parents and written parental consent to participate in the study (by the father if the mother is unable to participate)

Exclusion Criteria:

* Single parent or homosexual couple
* Absence of the father in the delivery room
* Parents not speaking French
* Skin temperature of the newborn < 36°C at the time of randomization
* Conditions not allowing the early skin-to-skin contact: omphalocele, gastroschisis, desquamating dermatological conditions (Harlequin syndrome, Collodion)
* Clinical condition requiring a specific transfer mode according to the pediatrician in the delivery room
* Parents under legal protection
* Minor parents

Ages: 24 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in the infant skin temperature due to the transfer procedure | During the transfer procedure
  Fluctuation in the infant skin temperature between the randomization in the delivery room and the admission in the neonatal intensive care unit (NICU)

SECONDARY OUTCOMES:
Change in the infant's heart rate during the transfer procedure | During the transfer procedure
  Heart rate values during the transfer procedure
Occurrence of bradycardia episodes in infant during the transfer procedure | During the transfer procedure
  Rapid decrease in heart rate less than 100 beats/min that lasts at least 10 secondes during the transfer procedure
Change in the infant's oxygen saturation during the transfer procedure | During the transfer procedure
  Oxygen saturation values during the transfer procedure
Occurrence of desaturation episodes in infant during the transfer procedure | During the transfer procedure
  Decrease in oxygen saturation less than 85% that last at least 10 secondes
Change in the infant's fraction of inspired oxygen during the transfer procedure | During the transfer procedure
  Fraction of inspired oxygen values during the transfer procedure
Duration of the transfer procedure | During the transfer procedure
  Time (in min) during the transfer procedure
First Hydrogen Potential (pH) of the newborn | First blood gas in the NICU
  First assessment of pH in the neonatal intensive care unit (NICU)
Carbon dioxide partial pressure (pCO2) of the newborn | First blood gas in the NICU
  First assessment of carbon dioxide partial pressure (pCO2) in the neonatal intensive care unit (NICU)
Blood glucose of the newborn | First blood glucose measurement in the NICU
  First assessment of blood glucose in the neonatal intensive care unit (NICU)
Occurence of hypothermia | From admission in the neonatal intensive care unit to 30 min later
  Decrease of skin temperature less than 36°C
Time to the first skin-to-skin contact in the neonatal care unit | Postnatal hour when the first skin-to-skin contact will occur in the neonatal care unit
  Postnatal hour when the first skin-to-skin contact will occur in the neonatal care unit
Practice of skin-to-skin contact in the neonatal intensive care unit (NICU) during the first week of life | During the first 7 days of the stay in the neonatal care unit
  Frequency of skin-to-skin contact (Postnatal day and hour), length of each skin-to-skin contact, which parent involves in each skin-to-skin contact episode.
Quality of parental bond | 2 time points: i) Between the infant postnatal day 3 and postnatal day 7, and ii) at the infant postnatal day 30 or at the end of the stay in the NICU if this event occur before the postnatal day 30
  Assessment through a maternal questionnaire: Mother-to-Infant Bonding Scale (MIBS) questionnaire (Mother-to-infant bonding scale - Taylor, 2005). Only the infant's mother will be invited to fill out this questionnaire.
Parental stress | 2 time points: i) Between the infant postnatal day 3 and postnatal day 7, and ii) at the infant postnatal day 30 or at the end of the stay in the NICU if this event occur before the postnatal day 30
  Parental stress assessed by Perceived Stress Scale (PSS) - Neonatal Intensive Care Unit (NICU) questionnaire (Perceived Stress Scale Neonatal Intensive Care Unit - Miles, 1993). The infant's mother and father will be invited to fill out this questionnaire.
Parental post-traumatic stress disorder | At the infant postnatal day 30 or at the end of the stay in the NICU if this event occur before the postnatal day 30
  Parental post-traumatic stress disorder assessed by Perinatal Post traumatic stress disorder Questionnaire (PPQ) - DEMIER, 1996). The infant's mother and father will be invited to fill out this questionnaire.
Infant growth: Weight | At birth and weight at the postmenstrual age of 36 weeks
  Weight at birth and at the postmenstrual age of 36 weeks
Infant growth: Height | At birth and at the postmenstrual age of 36 weeks
  Height at birth and at the postmenstrual age of 36 weeks
Infant growth: Head circumference | At birth and at the postmenstrual age of 36 weeks
  Head circumference at birth and at the postmenstrual age of 36 weeks
Neonatal morbidity and mortality at the postmenstrual age of 36 weeks | At the postmenstrual age of 36 weeks
  Death
  * Intraventricular hemorrhage (maximal grade),
  * Periventricular leukomalacia, Necrotizing enterocolitis (> stade 2 of the Bell classification),
  * Neonatal surgery,
  * Early onset sepsis (onset before postnatal day 2 and > 3 days of intravenous antibiotherapy),
  * Late onset sepsis (Blood culture positive, number of events),
  * Number of red blood cell transfusions,
  * Duration of mechanical ventilation (days).
  * Severe bronchopulmonary dysplasia,
  * Retinopathy of prematurity that requires laser photocoagulation or intravitreal injection of proangiogenic factor,
  * Length of stay in neonatal intensive care unit (days).
Modalities of breastfeeding | During the NICU stay: infant postnatal day
  First breastfeeding attempt in the neonatal intensive care unit (NICU)
Modalities of breastfeeding | At the postmenstrual age of 36 weeks
  Presence of complete or partial breastfeeding at the postmenstrual age of 36 weeks
Mode of infant feeding at the postmenstrual age of 36 weeks | At the postmenstrual age of 36 weeks
  Modes of infant feeding that include breastfeeding, breastmilk given through a bottle, artificial formula

OTHER OUTCOMES:
Self-questionnaires to study parents' experience of their infant hospitalization | 2 time points: i) Between the infant postnatal day 3 and postnatal day 7, and ii) at the infant postnatal day 30 or at the end of the stay in the NICU if this event occur before the postnatal day 30
  Ancillary study: Self-questionnaires to study parents' experience of their infant hospitalization to assess stress at different times.

CONTACTS AND LOCATIONS:
Overall Officials: Nolwenn CLENET, Study Director — University Hospital, Tours
Locations (5):
- France (5):
  - CHU Angers, Angers
  - Neonatal medicine and intensive care unit, University Hospital, Orléans, Orléans
  - Neonatal intensive care unit, University Hospital, Saint-Etienne, Saint-Etienne
  - Neonatology service, University Hospital, Toulouse, Toulouse
  - Neonatal and paediatric service, University Hospital, Tours, Tours